CLINICAL TRIAL: NCT06479590
Title: Investigate the Effects of Transcranial Direct Current Stimulation on Glucose Level in Healthy Young Adults: Crossover RCT
Brief Title: Effects of Transcranial Direct Current Stimulation on Glucose Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REC01893 Faryal Shoukat
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Glucose Metabolism Disorders
Keywords: tDCS; glucose uptake; healthy young
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS Group (Experimental)
  Interventions: Device: tDCS
- Sham Group (Sham Comparator)
  Interventions: Other: Sham tDCS

INTERVENTIONS:
Device: tDCS — The DCS electrode sheaths of 7x5 cm will be soaked with standard saline solution(NaCl 9%) and fixed by elastic bands. tDCS will deliver 20 min of anodal stimulation (1-2mA, fade in/out 8 sec)
  Arms: tDCS Group
Other: Sham tDCS — sham-tDCS will be applied for 30 s to make it difficult for the individual to distinguish the placebo from a real tDCS application
  Arms: Sham Group

SUMMARY:
Previous studies have investigated the impact of tDCS on systemic glucose, neglecting to explore its effects on diabetic factors and its safety. Some studies used small sample size, limiting the ability to identify significant impacts or generalized findings to large population.

DETAILED DESCRIPTION:
The proposed study suggests addressing these gaps by employing a large sample size, comprehensive outcome measurements, assessing tDCS impact on diabetes mellitus (DM) risk variables, and integrating ethical considerations into the research design and implementation. The study aims to fill existing gaps in knowledge about tDCS effects on blood glucose regulation and diabetic risk factors by conducting more robust research methodologies The effects of tDCS on addictive behavior and cerebral glucose metabolism in problematic online gamers were examined in a single-blinded RCT. Over a 4-weekperiod, participants received 12 sessions of either active or sham tDCS to the dorsolateral prefrontal cortex. In the active group, glucose metabolism was enhanced in certain brain regions, showing decreased addiction severity in both groups. As a result of these findings, it appears that prefrontal tDCS is capable of controlling gaming behaviors and enhancing cerebral glucose metabolism

ELIGIBILITY:
Inclusion Criteria:

* Both Male & Female
* Age 18-30 years

Exclusion Criteria:

* Pregnancy
* Lactating mothers
* Skin Irritation and Allergies
* Brain Tumor or Shunt
* Brain Metallic implants
* Epileptic disease
* GI Disorder and Endocrine Disorder
* Drug abuse
* History of medications any hormonal therapy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
RBS | 2-4 hours
  Two hours after meal, peripheral venous blood samples are collected to check random blood glucose levels. The morning random glucose level had a linear relationship with glycated haemoglobin levels taken simultaneously. A blood glucose level of 7 mmol/l had 92.7% sensitivity for good control (HbA1c < or = 7.8%) on a blood sample which was taken simultaneouslyand59.8% specific for the same
6 Minute walk test | baseline
  The 6-minute walk test (6MWT) is widely employed in clinical settings due to its ease of administration, good tolerance, and safety. It assesses functional exercise capacity by measuring the distance an individual walks in 6 minutes. Moreover, it serves as a valuable predictor of morbidity and mortality across various cardiopulmonary conditions, demonstrating excellent reliability (ICC = 0.9) and validity in healthy adults.

SECONDARY OUTCOMES:
International physical activity questionnaire (IPAQ-SF) | baseline
  This cost-effective measure will assess participants' physical activity intensity and sitting time to estimate total physical activity in MET-min/week. It records activity levels across four categories: vigorous-intensity (e.g., aerobics), moderate-intensity (e.g., leisure cycling), walking, and sitting. The International Physical Activity Questionnaire Short Form(IPAQ-SF)demonstrates good test-retest reliability (ICC > 0.65) and satisfactory criterionvalidity in healthy adults
Rapid Assessment of Physical Activity (RAPA) | baseline
  RAPA is a self-administered questionnaire comprising 9 items with yes or no responses, determining the level of physical activity. The first 7 items assess aerobic activity (RAPA 1), while the last 2 items focus on strength and flexibility(RAPA 2) and are not included in the total score. Test-retest reliability for RAPA in healthy adults is high, with a calculated value of 0.996 (95%CI0.992-0.998), indicating very good reliability
Finish Diabetes Risk Score | baseline
  The Finnish Diabetes Risk Score (FINDRISC) questionnaire is a validated tool for predicting type 2 diabetes risk. It estimates the probability of developing diabetes within the next 10 years. FINDRISC demonstrates excellent reliability, with an Intra class Correlation Coefficient (ICC) of 0.94.
GAD-7 | baseline
  The 7-item Generalized Anxiety Disorder Scale (GAD-7) is a self report tool for assessing symptoms of GAD, including excessive and uncontrollable anxiety and worry lasting at least 6 months. The scale demonstrates excellent reliability in young adults, with a cronbach'sαcoefficient of 0.895, surpassing the recommended threshold of 0.80
Waist and Hip Ratio | baseline
  Waist and hip circumference measurements serve as cost-effective, non-invasive indicators of body fat distribution and disease risk. High Intra class Correlations (ICC) between self and technician measurements are observed, with values of 0.97 for waist and 0.96 for hip circumference. Additionally, self-measurements at home exhibit high test-retest reliability, with ICC values of at least 0.87 when compared to lab measurements
BMI | baseline
  Body Mass Index (BMI) is a measure utilizing height and weight to assess obesity, with values ranging from <18.5 to >30. BMI demonstrates high reliability, with an Intra class Correlation Coefficient (ICC) of 0.96

CONTACTS AND LOCATIONS:
Overall Officials: Sumaiyah Obaid, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kraus C, Hahn A, Sigurdardottir H, Spurny B, Wadsak W, Mitterhauser M, Hacker M, Kasper S, Lanzenberger R. Brain glucose uptake during transcranial direct current stimulation measured with functional [18F]FDG-PET. Brain Imaging Behav. 2020 Apr;14(2):477-484. doi: 10.1007/s11682-019-00195-4. PMID 31598826
- [Background] Kistenmacher A, Manneck S, Wardzinski EK, Martens JC, Gohla G, Melchert UH, Jauch-Chara K, Oltmanns KM. Persistent blood glucose reduction upon repeated transcranial electric stimulation in men. Brain Stimul. 2017 Jul-Aug;10(4):780-786. doi: 10.1016/j.brs.2017.03.011. Epub 2017 Mar 25. PMID 28392373
- [Background] Binkofski F, Loebig M, Jauch-Chara K, Bergmann S, Melchert UH, Scholand-Engler HG, Schweiger U, Pellerin L, Oltmanns KM. Brain energy consumption induced by electrical stimulation promotes systemic glucose uptake. Biol Psychiatry. 2011 Oct 1;70(7):690-5. doi: 10.1016/j.biopsych.2011.05.009. Epub 2011 Jun 24. PMID 21703596